CLINICAL TRIAL: NCT02967627
Title: Incisional Negative Pressure Wound Therapy Following Colorectal Resection: a Single Site, Prospective, Randomized Control Trial
Brief Title: VAC Dressings for Colorectal Resections
Acronym: VACCRR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-02565
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Surgical Site Infection; Wound Complication; Wound Dehiscence; Seroma; Hematoma
MeSH Terms: conditions — Surgical Wound Infection; Seroma; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incisional Negative Pressure Wound Therapy (iNPWT) (Experimental): Patients in the iNPWT group will have their incision covered by a single layer of Mepitel wound contact layer followed by application of a KCI V.A.C Simplace ™ Dressing composed of a strip of black foam covering the entire length of the incision followed by coverage of the incision, Mepitel, and foam with an occlusive Tegederm ™ dressing to establish an airtight seal. Negative pressure will then be applied using a SensaT.R.A.C. Pad ™ to a setting of 100 mmHg continuous suction. Dressings shall remain in place and will be removed by the surgical team on the morning of the third post-operative day and left open to air thereafter. Any loss of seal of the dressing shall be reinforced using occlusive dressings.
  Interventions: Device: Incisional Negative Pressure Wound Therapy (iNPWT)
- Standard Therapy (Active Comparator): Patients in the conventional dressings group will receive a standard Mepore ™ dressing applied to cover the entire incision. This will be left in place and and removed by the surgical team on the morning of the second postoperative day and will be left open to air thereafter. Dressings may be either reinforced or changed at the discretion of the surgical team due to drainage or saturation during the first two postoperative days.
  Interventions: Device: Sterile Gauze Dressing

INTERVENTIONS:
Device: Incisional Negative Pressure Wound Therapy (iNPWT) — Incisional Negative Pressure Wound Therapy devices are lightweight, self contained, portable battery powered (or line powered), suction pumps for medical procedures where secretions and other body fluids and infectious materials must be removed through the application of continuous or intermittent negative pressure. The pumps are operated through computer software, having help and alarm features. The device is indicted for management of chronic, acute, traumatic, subacute and dehisced wounds, partial-thickness burns, ulcers (such as diabetic or pressure), flaps and grafts. The pumps may be used at patient's bedside. These are suitable for use in either hospitals or long term care facilities and nursing homes. These devices will be applied to closed laparotomy incisions with the aim to provide three days of continuous negative pressure of - 100mmHg.
  Other Names: Surgical Incision Management System (SIMS); Closed Incisional Negative Pressure Wound Therapy (ciNPWT); V.A.C dressing
  Arms: Incisional Negative Pressure Wound Therapy (iNPWT)
Device: Sterile Gauze Dressing — In most cases, self-adhesive, absorbent dressings will be used for standard wound therapy. However, surgical teams may decide on alternative forms of sterile gauze dressings, as long as the wound site is kept clean and dry. Dressings should be taken down on the second post-operative day.
  Other Names: Self-adhesive Absorbent Dressing
  Arms: Standard Therapy

SUMMARY:
Surgical Site Infections (SSIs) and wound complications are common occurrences following colorectal resection surgery. Incisional Negative Pressure Wound Therapy (iNPWT) has developing evidence for improving wound complication rates in certain populations. However, there have been no RCTs to date that have looked at iNPWT use after colorectal surgery. We propose a study in which patients are randomized into one of two treatment arms: 1) incisional NPWT, and 2) standard sterile gauze dressings. Patients will be followed for 30 days for diagnosis of infection or wound complication. We will compare primary outcomes in each group using Chi-Squared statistical testing in order to report a Absolute Risk Reduction and Number Needed to Treat

DETAILED DESCRIPTION:
Purpose: To evaluate if incisional Negative Pressure Wound Therapy (iNPWT) confers a lower rate of Surgical Site Infection (SSI) or wound complication compared to standard treatment of elective colorectal resection laparotomies.

Justification: Colorectal resection with bowel anastomosis is a clean-contaminated procedure known to have increased rates wound complication. Techniques like the use of incisional wound barriers, antimicrobial eluding dressings or iodine washout have been assessed in an attempt to reduce occurrence. However, evidence for their efficacy is not compelling for surgeons to universally adapt. Meanwhile, negative pressure wound therapy has demonstrated impressive efficacy in the management of complex and non-healing wounds. And recently, NPWT has become an area of interest in managing, not only open wounds, but closed wounds as well. The benefit of this therapy is yet to be clearly defined in the elective colorectal resection patient population, however.

Null hypothesis: There is no difference in SSI or wound complication rate in standard and iNPWT groups.

Design: Single-institution, prospective, randomized, open-label, superiority trial

Statistical Analysis: Assuming a complication rate of 20-30% and a relative risk reduction of 50%, we will recruit 400 patients (200 in each group) to achieve a power of 80% and type 1 error of 0.05. Primary endpoints will be: Wound Complication - defined as presence of seroma, hematoma, dehiscence, SSI - and SSI reported independently. Secondary endpoints will include: Length of Stay, ER visits related to SSI, Complications (according to Clavien-Dindo classification), need for and duration of home care related to wound care, and wound VAC specific complications (local reaction to adhesive dressing, blisters, failure of vacuum, need for early removal). Primary endpoints will be assessed according to intention-to-treat principle using Pearson's chi-squared test. In the event that baseline characteristics are significantly different, a secondary analysis using multivariable logistic regression will adjust for the effect of the difference. A p value of < 0.05 will be used to determine significance. Results will be presented as an absolute risk reduction as well as number needed to treat to prevent one wound complication. Secondary outcomes will be compared using a Mann-Whitney U-test for non-normally distributed continuous variables and chi-squared for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* elective colorectal resection for benign or malignant disease
* surgery involves an anastomosis
* open or minimally invasive technique
* midline laparotomy used for specimen extraction

Exclusion Criteria:

* under 19
* allergy/sensitivity to adhesives
* immunocompromised
* pregnant
* emergency surgery
* elective surgery
* additional procedures performed at time of surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Superficial Surgical Site Infection (SSI) | 30 days post op
  Infection occurring within the first thirty days after surgery with at least one of the following: 1) purulent drainage from the superficial incision; 2) organisms obtained from an aseptically obtained culture of tissue or fluid from the superficial incision; 3) at least one of the local signs of infection; 4) superficial incision deliberately opened by the surgeon (unless the culture is negative)
Wound Complication | 30 days post op
  At least one of the following: 1) seroma; 2) hematoma; 3) SSI; 4) wound dehiscence/disruption

SECONDARY OUTCOMES:
Length of stay | approximately 5-10 days on average
  Number of days spent in hospital post op
Wound-related visits post surgery | 30 days post op
  Number of wound-related visits to primary care physician, nurse practitioner, or emergency for concerns related to laparotomy incision.
Need for and duration of home care | 30 days post op
  Did the patient require home care nursing for wound care? If so, how many visits?
Blistering/reaction to wound dressings | 3 days post op
  Did the patient develop skin blisters or hypersensitivity reaction secondary to their wound dressings?
Post Op Complications | 30 days post op
  Did the patient develop any major complications - as according to Clavien-Dindo classification?

CONTACTS AND LOCATIONS:
Overall Officials: Neely O.M. Panton, MD, FRCSC, Principal Investigator — UBC Division of General Surgery

IPD SHARING:
Plan to Share IPD: Undecided
To be decided